CLINICAL TRIAL: NCT01963494
Title: Days in Motion: A Planning Intervention Study With Couples to Enhance Daily Physical Activity (DiM)
Brief Title: Days in Motion: A Planning Intervention Study With Couples to Enhance Daily Physical Activity
Acronym: DiM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Freie Universität Berlin (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Principal Investigator, Nina Knoll, Univ.-Prof. Dr. Nina Knoll, Freie Universität Berlin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110014
Record Dates: First submitted 2013-09-30; First posted 2013-10-16 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Health Behavior; Physical Activity; Couples
Keywords: Physical activity; Health-behavior-change; Dyadic Planning; Individual Planning
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dyadic planning intervention (Experimental): A general motivational treatment is provided to each participant. For randomly assigned couples, randomly selected target persons form action plans to increase daily physical activity together with their partners.
  Interventions: Behavioral: Dyadic planning intervention; Behavioral: General motivational treatment
- Individual planning intervention (Active Comparator): A general motivational treatment is provided to each participant. For randomly assigned couples, target persons form action plans individually to increase daily physical activity and partners receive a distraction task.
  Interventions: Behavioral: Individual planning intervention; Behavioral: General motivational treatment
- No-planning control condition (Active Comparator): A general motivational treatment is provided to each participant. For randomly assigned couples, target persons do not receive instructions for action planning, but perform a distraction task together with their partners.
  Interventions: Behavioral: General motivational treatment

INTERVENTIONS:
Behavioral: Dyadic planning intervention — Dyadic planning refers to creating together with a partner if-then plans on when, where, and how the individual target person will implement a new behaviour.
  Arms: Dyadic planning intervention
Behavioral: Individual planning intervention — Target persons form action plans on their own.
  Arms: Individual planning intervention
Behavioral: General motivational treatment — Both partners are asked to read a brochure that aims at enhancing their motivation to increase levels of moderate physical activity. They respond to a quiz afterwards.

SUMMARY:
Regular physical activity is one prominent health-protective behaviour which might increase with the help of self-regulatory strategies such as action planning.

The aim of this randomised controlled trial is to examine changes in daily moderate physical activity in couples following (a) a dyadic planning intervention, (b) an individual planning intervention or (c) a no-planning control condition. Changes in daily physical activity will be examined over a period of one year.

It is assumed that target persons from couples receiving a dyadic planning intervention will show greater increases in daily physical activity than target persons from couples receiving an individual planning intervention. For couples receiving a dyadic planning intervention or an individual planning intervention, it is hypothesized that target persons will show higher increases in daily physical activity than target persons from couples participating in the no-planning control condition.

DETAILED DESCRIPTION:
Regular physical activity reduces the risk of a number of grave chronic diseases, including many forms of cancer. Guidelines indicate that increasing moderate physical activity by 30 to 60 minutes on at least 5 days of the week should already be associated with such significant health benefits. However, recent epidemiologic information indicates that only about 20% of the German adult population fully meet this important health behaviour goal.

Despite this relatively moderate recommended increase in physical activity and an apparently high acceptance of goals to increase moderate daily physical activity, many people fall short of goal achievement, as the implementation and maintenance of behaviour change often fails. Therefore, aside from enhancing motivational factors, interventions promoting health-behaviour change (e.g., increase in physical activity), are now commonly extended to address volitional strategies, such as action planning. Action planning aids individuals in translating their goals into behaviour. By forming action plans, individuals link situational cues ('when' and 'where' specifications of critical situations) to behavioural responses ('what to do' or 'how to act') in an 'if-then'-format. Available findings suggest that action planning aside from its direct effects on behaviour change, including increase in physical activity, also fosters other self-regulation strategies that are effective in the implementation and maintenance of changes in health-related behaviour. Research on action planning so far mainly focuses on its benefits for the individual's self-regulation of behaviour. To date there is little evidence on the role of the close social environment in planning health-behaviour change. However, married and cohabiting individuals often try to and succeed in coregulating their partners' health behaviour, including partners' levels of physical activity. Therefore, in the proposed study, an extension of individual action planning to the level of the dyad, i.e., dyadic planning, will be examined, along with associated mechanisms fit to aid the process of increasing physical activity. Dyadic planning refers to creating together with a partner if-then plans on when, where and how the individual target person will implement a new behaviour (e.g., be more physically active). We hypothesise that dyadic planning leads to higher increases in daily physical activity when compared to individual planning or no planning.

In the proposed randomised controlled trial, we will compare changes in daily moderate physical activity in N = 346 adults (primary outcome) and their partners who receive a general motivational treatment to enhance daily physical activity and are then randomly assigned to one of three intervention conditions: (a) a dyadic planning intervention, in which target persons form action plans to increase daily physical activity together with their partners, or (b) an individual planning intervention, in which target persons form such action plans individually and partners receive a distraction task, or (c) a no-planning control condition, in which target persons do not receive instructions for action planning, but perform a distraction task together with their partners. The study will entail an experimental longitudinal design with a baseline assessment (T0), an intervention session one week following baseline (T1) and follow-up assessments at 1 week (T2), 6 (T3; primary endpoint), 19 (T4), 26 (T6), and 52 (T7) weeks following the main intervention session. A booster intervention (T5) will take place 20 weeks after the main intervention session, i.e. 1 week following T4. Objective measurement of daily physical activity will include 4 one-week (T0, T2, T3, T7) accelerometer assessments. Additionally, further objective measurements of cardiorespiratory fitness, BMI, and waist-to-hip ratios along with self-report assessments from target persons and partners will be collected. Proposed mechanisms of the total intervention effect along with covariates will be assessed mostly via self-report.

Results of this study will contribute to the still limited understanding of the interplay of individual and dyadic regulation in the increase of daily physical activity and its maintenance, both in persons targeted by the intervention and in their partners. Findings will guide further development of this economical dyadic planning intervention that can be straightforwardly implemented in clinical settings to support the initiation and maintenance of preventive behaviour in couples. Furthermore, this theoretically-derived dyadic planning intervention can easily be extended to other domains of health-behaviour change.

ELIGIBILITY:
Inclusion Criteria:

* Married and/or cohabiting couples who are currently in a romantic relationship and have been living together for a minimum of 6 months

Exclusion Criteria:

* Being a minor (i.e., younger than 18 years)
* Restrictions on being physically active as assessed by a risk-check form modelled after the Physical Activity Readiness Questionnaire
* Being a competitive athlete and engaging in vigorous physical exercise for more than 3 hours per day
* Participating in other intervention programmes targeting physical activity or weight-loss
* Self-reported severe cardio-vascular or pulmonary disease, diseases or injury of the musculoskeletal system, degenerative neurological diseases, paraplegia
* Pregnancy
* A BMI below 17.5
* Insufficient comprehension of the German language

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2013-03; Primary Completion 2015-02 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Physical activity | six weeks post intervention
  Target persons' change in moderate daily physical activity (in minutes) from baseline (T0) until 6-weeks (T3) following the intervention will be assessed by an accelerometer device. At each assessment, accelerometer devices will be worn for 7 days.

SECONDARY OUTCOMES:
Cardiorespiratory fitness | one year post intervention
  Cardiorespiratory fitness in target persons and partners is measured by a 2-km walking test. Using the duration and heart-rate of the 2-km walking test, as well as age, sex and BMI, an index is calculated that represents the cardiorespiratory fitness measure which can be compared to norm values.
Dyadic action planning | one year post intervention
  Dyadic action planning of daily physical activity will be assessed in target persons and partners by questionnaire.
  Couples' own regular dyadic action planning of target persons' and partners' daily physical activity during the past seven days will be assessed by four items using the stem "I have made a detailed plan together with my partner regarding ..." followed by (1) "when", (2) "where", (3) "how", and (4) "how often to be physically active" adapted from earlier research on dyadic planning of pelvic-floor training (Burkert et al., 2011). Response options range from 1 = "does not apply at all" to 6 = "applies exactly".
Individual action planning | one year post intervention
  Individual action planning of daily physical activity will be assessed in target persons and partners by questionnaire.
  Participants' own regular individual action planning of daily physical activities during the past seven days will be measured using four items using the stem "I have made a detailed plan regarding ..." followed by (1) "when", (2) "where", (3) "how", and (4) "how often to be physically active" (Scholz et al., 2007). Response options range from 1 = "does not apply at all" to 6 = "applies exactly".
Physical activity | one year post intervention
  Partners' daily physical activity will be objectively assessed in a parallel manner at the same four measurement occasions (T0, T2, T3, and T7). At each assessment, accelerometer devices will be worn for 7 days. Accelerometers will be worn by target persons and partners, providing data on activity counts, steps taken, activity intensity levels, and METs.
Physical activity | one year post intervention
  Self-reported physical activity in target persons and partners is assessed by a combination of the Office in Motion questionnaire (OIMQ; Mäder et al., 2006) complemented by items of the Physical Activity Frequency Questionnaire (PAFQ; Bernstein, Sloutiskis, Kumanyika, Sparti, Schutz, & Morabia, 1998). This combined measure provides detailed information on time spent on physical activities of moderate and vigorous intensity within the past 7 days, covering the domains of transportation, occupational activity, household and yard work activities, and leisure-time physical activity.
Individual action control | one year post intervention
  Physical activity-related individual action control during the past seven days will be assessed by 6 items addressing the three action control facets of comparative self-monitoring, awareness of standards, and self-regulatory effort (e.g., "During the last seven days I have really tried to be regularly physically active"; Sniehotta et al., 2005). Response options range from 1 = "does not apply at all" to 6 = "applies exactly".
Received partner support | one year post intervention
  Physical activity-related received partner support during the past seven days will be assessed using 6 items from the Berlin Social Support Scales (Schulz & Schwarzer, 2004) adapted to the domain of physical activity (e.g., "My partner helped me to be physically active"). Response options range from 1 = "does not apply at all" to 6 = "applies exactly".
Provided partner support | one year post intervention
  Physical activity-related provided partner support during the past seven days will be assessed using 6 items from the Berlin Social Support Scales (Schulz & Schwarzer, 2004) adapted to the domain of physical activity. These items will mirror the received support items (e.g., "I helped my partner to be physically active"). Response options range from 1 = "does not apply at all" to 6 = applies exactly".
Received partner control | one year post intervention
  Physical activity-related received partner control during the past seven days will be assessed with a measure adapted from Lewis and Rook (1999). The scale consists of 8 items (e.g., "My partner pressured me to be physically active") measuring received partner control related to physical activity. Response options range from 1 = "does not apply at all" to 6 = "applies exactly".
Provided partner control | one year post intervention
  Physical activity-related provided partner control during the past seven days will be assessed in accordance with Lewis and Rook (1999) by 8 items (e.g., "I pressured my partner to be physically active") applied to physical activity. Response options range from 1 = "does not apply at all" to 6 = "applies exactly".

CONTACTS AND LOCATIONS:
Overall Officials: Nina Knoll, Univ.-Prof., Study Chair — Freie Universität Berlin
Locations (1):
- Freie Universität Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Burkert S, Scholz U, Gralla O, Roigas J, Knoll N. Dyadic planning of health-behavior change after prostatectomy: a randomized-controlled planning intervention. Soc Sci Med. 2011 Sep;73(5):783-92. doi: 10.1016/j.socscimed.2011.06.016. Epub 2011 Jul 12. PMID 21807446
- [Background] Scholz U, Sniehotta FF, Burkert S, Schwarzer R. Increasing physical exercise levels: age-specific benefits of planning. J Aging Health. 2007 Oct;19(5):851-66. doi: 10.1177/0898264307305207. PMID 17827449
- [Background] Bernstein M, Sloutskis D, Kumanyika S, Sparti A, Schutz Y, Morabia A. Data-based approach for developing a physical activity frequency questionnaire. Am J Epidemiol. 1998 Jan 15;147(2):147-54. doi: 10.1093/oxfordjournals.aje.a009427. PMID 9457004
- [Background] Mader U, Martin BW, Schutz Y, Marti B. Validity of four short physical activity questionnaires in middle-aged persons. Med Sci Sports Exerc. 2006 Jul;38(7):1255-66. doi: 10.1249/01.mss.0000227310.18902.28. PMID 16826022
- [Background] Sniehotta, F. F., Scholz, U., & Schwarzer, R. (2005). Bridging the intention-behaviour gap: Planning, selfefficacy, and action control in the adoption and maintenance of physical exercise. Psychology & Health, 20, 143-160.
- [Background] Schulz, U., & Schwarzer, R. (2004). Long-term effects of spousal support on coping with cancer after surgery. Journal of Social and Clinical Psychology, 23, 716-732.
- [Background] Lewis MA, Rook KS. Social control in personal relationships: impact on health behaviors and psychological distress. Health Psychol. 1999 Jan;18(1):63-71. doi: 10.1037//0278-6133.18.1.63. PMID 9925047
- [Derived] Knoll N, Hohl DH, Keller J, Schuez N, Luszczynska A, Burkert S. Effects of dyadic planning on physical activity in couples: A randomized controlled trial. Health Psychol. 2017 Jan;36(1):8-20. doi: 10.1037/hea0000423. Epub 2016 Sep 19. PMID 27642760
- See also: Related Info — http://www.ewi-psy.fu-berlin.de/einrichtungen/arbeitsbereiche/gesund/forschung/bewegter_alltag